CLINICAL TRIAL: NCT04009226
Title: International GNE Myopathy Patient Registry (GNE001)
Brief Title: International GNE Myopathy Patient Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 13/NE/0123
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2019-07

CONDITIONS: GNE Myopathy; Hereditary Inclusion Body Myopathy
Keywords: Distal Myopathies; Neuromuscular Diseases; Muscular Dystrophies; GNE Myopathy; Hereditary Inclusion Body Myopathy
MeSH Terms: conditions — Distal myopathy, Nonaka type; Distal Myopathies; Neuromuscular Diseases; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with GNE
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Participants who have volunteered to participate will complete various questionnaires relating to their condition.

SUMMARY:
GNE myopathy, an ultra-rare disease, is a severe progressive myopathy that typically presents in early adulthood as weakness in the distal muscles of the lower extremities and progresses proximally, leading to a loss of muscle strength and function, and ultimately a wheelchair-bound state. The rate of progression is gradual and variable over the course of 10-20 years or longer.

There is a need to understand the world wide epidemiology of this ultra-rare condition, better understand a long-term disease course and the progression of disease-specific features, support translational research by evaluating burden illness and support clinical research recruitment. Therefore, the study will longitudinally collect information via an online patient registry platform.

DETAILED DESCRIPTION:
GNE myopathy is an ultra- rare condition. Most of the knowledge is coming from case reports or small cohort observations. There is a need to more precisely understand the long-term disease course and the progression of disease-specific features of GNE myopathy, and in turn characterise the overall burden of this illness. Also, to better understand the disease, describe it variability, genotype-phenotype correlation, quality of life, epidemiology, health-economics aspects and need for assistive walking devices. Collected data needs to be harmonised to be compatible collaborative work with Remudy (Japanese patient registry). This collaborative effort will enable the analysis of the largest GNE myopathy data set in the world. To this end, this study will collect patient information longitudinally. Upon patient's agreement, the registry curator can contact nominated clinicians to request additional data or data validation.

Study Objectives

The objectives of the study are to:

* Longitudinally characterize disease-specific features of GNE myopathy
* Characterize the burden of illness and quality of life in patients with GNE myopathy
* Support recruitment in research activities
* Inform registry participants via newsletters about scientific developments in the GNE myopathy field

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at the time of informed consent
* Clinical and/or genetic diagnosis of GNE myopathy (also known as HIBM, QSM, Inclusion Body Myopathy Type 2, DMRV, or Nonaka disease)
* Willing and able to provided electronic (or written) consent and comply with all study requirements.

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must have a diagnosis of GNE myopathy (also known as HIBM, Quadriceps Sparing Myopathy (QSM), Inclusion Body Myopathy Type 2, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease)
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Disease history | 12 months
  Patient reported disease history including GNE myopathy diagnosis.
General medical history | 12 months
  Patient reported general medical history.
Medication use | 12 months
  Patient reported medical use.
Quality of life questionnaire (non-validated) | 12 months
  Patient reported quality of life
Level of physical activity | 12 months
  Patient reported level of physical activity
Muscle biopsy and genetic testing status | 12 months
  Patient reported history of muscle biopsy and details of whether they have undergone genetic testing for GNE myopathy

CONTACTS AND LOCATIONS:
Overall Officials: Volker Straub, MD, PhD, Principal Investigator — John Walton Muscular Dystrophy Research Centre
Locations (1):
- John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne, United Kingdom